CLINICAL TRIAL: NCT06818396
Title: Analgesic Efficacy of Fascia Iliaca Compartment Block Compared With Intrathecal Nalbuphine for Hip Surgery Under Spinal Anesthesia: a Randomized Controlled Trial
Brief Title: Analgesic Efficacy of Fascia Iliaca Compartment Block Compared With Intrathecal Nalbuphine for Hip Surgery Under Spinal Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ibrahim Mamdouh Esmat, Professor of Anesthesia and Intensive Care,Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU-MS 72 / 2025
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- US-guided fascia iliaca compartment block (FICB) and spinal anesthesia (Active Comparator)
  Interventions: Other: US-guided fascia iliaca compartment block (FICB) and spinal anesthesia
- Intrathecal nalbuphine and spinal anesthesia (Active Comparator)
  Interventions: Drug: Intrathecal nalbuphine and spinal anesthesia
- Spinal anesthesia (Other)
  Interventions: Other: Spinal anesthesia

INTERVENTIONS:
Other: US-guided fascia iliaca compartment block (FICB) and spinal anesthesia — US-guided fascia iliaca compartment block (FICB) and spinal anesthesia
  Arms: US-guided fascia iliaca compartment block (FICB) and spinal anesthesia
Drug: Intrathecal nalbuphine and spinal anesthesia — intrathecal nalbuphine and spinal anesthesia
  Arms: Intrathecal nalbuphine and spinal anesthesia
Other: Spinal anesthesia — Spinal anesthesia
  Arms: Spinal anesthesia

SUMMARY:
It is already known that fascia iliaca compartment block and intrathecal nalbuphine are very effective ways in postoperative pain control in patients having hip surgeries.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) score (ASA I- ASA II).
* Age ≥ 21years.
* Body mass index < 35 kg/m2

Exclusion Criteria:

* Patient's refusal.
* Known coagulopathy.
* Known peripheral neuropathy or neurological deficits.
* Known allergy to study drugs

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Time to first rescue analgesia (minutes). | in the first 24 hours after surgery
  Time to first rescue analgesia (minutes).

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University Hospitals, Cairo, Egypt